CLINICAL TRIAL: NCT05616702
Title: Effectiveness of Pressure Biofeedback Therapy and Progressive Muscle Relaxation Technique in Improving Pain and Disability Among Patients With Non-Specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Shaiaza Masooma, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2694
Record Dates: First submitted 2022-10-29; First posted 2022-11-15 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain, Mechanical; Chronic Low-back Pain; Mechanical Low Back Pain; Lower Back Pain Chronic; Low Back Pain; CLBP - Chronic Low Back Pain; Pain, Chronic; Pain, Back
Keywords: Pressure Biofeedback therapy; progressive muscles relaxation technique; chronic non-specific low back pain; chronic low back pain; non specific back pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Back Pain | interventions — Hyperthermia, Induced

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pressure Biofeedback Therapy + Progressive Muscle Relaxation Technique + Thermotherapy. (Experimental): This study ARM will receive following therapies
  1. Pressure Biofeedback Therapy
  2. Progressive Muscles Relaxation Technique
  3. Thermotherapy
  Interventions: Other: Pressure Biofeedback Therapy + Progressive Muscles Relaxation + thermotherapy
- Progressive Muscle Relaxation Technique + Thermotherapy (Active Comparator): This study ARM will receive following therapies
  1. Progressive Muscles Relaxation Technique
  2. Thermotherapy
  Interventions: Other: Progressive Muscles Relaxation + thermotherapy

INTERVENTIONS:
Other: Pressure Biofeedback Therapy + Progressive Muscles Relaxation + thermotherapy — Pressure Biofeedback Therapy
  * prone position, abdominal drawing in for 10 sec. (PBU inflated to 70 mmHg)
  * Supine position with flexed knees, abdominal drawing in for 10 sec. (PBU inflated to 40 mmHg)
  * Progress to leg loading in supine abdominal drawing in for 10 sec. (PBU inflated to 40 mmHg)
  Exercising dosage:
  * Duration: 15 mins
  * Frequency: 3 sessions/ week
  * Repetitions: 3 sets of 15 reps
  Progressive Muscles Relaxation Technique
  * Tense => five seconds and,
  * release => ten seconds (Each group of muscle)
  * 2 circuits daily
  Exercising dosage:
  * Duration: 15 mins
  * Frequency: weekly 3 sessions; for 6 weeks
  * Repetitions: 2 reps (cycles)
  Thermotherapy at lumbar region via electrical heating pad Duration: 15 mins
  Arms: Pressure Biofeedback Therapy + Progressive Muscle Relaxation Technique + Thermotherapy.
Other: Progressive Muscles Relaxation + thermotherapy — Progressive Muscles Relaxation Technique
  * Tense => five seconds and,
  * release => ten seconds (Each group of muscle)
  * 2 circuits daily
  Exercising dosage:
  * Duration: 15 mins
  * Frequency: weekly 3 sessions; for 6 weeks
  * Repetitions: 2 reps (cycles)
  Thermotherapy at lumbar region via electrical heating pad Duration: 15 mins
  Arms: Progressive Muscle Relaxation Technique + Thermotherapy

SUMMARY:
Low back pain is common MSK disease with prevalence of 60 to 70 percent. Patients with low back discomfort are typically treated conservatively by physical therapists. Progressive muscles relaxation technique has been shown in several studies to reduce chronic back pain and increase flexibility. pressure biofeedback therapy works on Intra abdominal pressure.it helps to alleviate compression on lumbar spine and support the adjacent lumbar spine.The aim of this randomized controlled trial is to determine the effectiveness of pressure biofeedback training (Pr.BFB) in combination with progressive muscles relaxation technique (PMR) & progressive muscles relaxation training alone on pain, disability, ROM & endurance of muscles among nonspecific chronic low back pain patients.

DETAILED DESCRIPTION:
A randomized clinical trial will be carried out in the Physical Therapy O.P.D of Dow hospital Karachi. Collection of data will commence right after approval of synopsis from Dow IRB. A sample of 70 NSCLBP patients calculated by using mean & SD of visual analogue scale in abdominal stabilisation training with Pr.BFB stabilizer was 2.69 ±0.93 and Progressive muscular Relaxation VAS was 3.863 ±2.03. Before being recruited into the experiment, patients will be screened to ensure that they meet the inclusion criteria. Pain rating scale and Roland-Morris questionnaire will be used to gather data after explaining the research goals to patients and obtaining formal consent from them. Patients will be divided into 2 interventional groups by simple random sampling, with 35 patients in each group. Experimental group will be received Pressure Bio-Feedback Therapy in combination with PMR Technique and Thermotherapy. The Control group, on the other hand, will be received a combination of Progressive Muscle Relaxation Technique and Thermotherapy for non-specific CLBP. It will be a 6-weeks intervention plan with 3 sessions per week (40-minutes each). Assessor will be blinded to the treatment. Roland Morris Low back pain and disability questionnaire (RMQ) and the NPR Scale will be used as primary outcome measures. Secondary outcomes will be determined by modified-modified Schober test for assessing lumbar ROM & Pressure Biofeedback Stabilizer unit helps to gauge muscular endurance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and referred patients with non-specific low back pain for more than 3 months
* 30 to 50 years
* Both genders

Exclusion Criteria:

* Any surgical history of lumbar spine
* Infections of the spine, malignancy
* Disc protrusion
* History of spinal fractures

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-10-16 (Estimated); Study Completion 2023-11-27 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (change is being assessed) | Baseline and 6 weeks
  On a scale of 0 to 10, "Please indicate the intensity of current, best, and worst pain levels over the past 24 hours on a scale of 0 (no pain) to 10 (worst pain imaginable)"
Roland-Morris Low Back Pain and Disability Questionnaire (change is being assessed) | Baseline and 6 weeks
  A standard tool called the "Roland-Morris Disability Questionnaire" consists of 24 items about a person's disabilities and pain perceptions The patient is told to draw a mark beside each element that corresponds to him or her. Sum of marked items will determine a patient's score. The scoring ranges from 0 - 24. (No to extreme disability).

SECONDARY OUTCOMES:
Endurance test (change is being assessed) (mmHg) | Baseline and 6 weeks
  For evaluating the functionality of deep abdominals via Pressure Biofeedback Unit , a standard device that monitors changes in pressure, allowing for muscle contraction and detection of spinal mobility during exercise.
Endurance test (change is being assessed) (hold time in seconds) | Baseline and 6 weeks
  For evaluating the functionality of deep abdominals via Pressure Biofeedback Unit , a standard device that monitors changes in pressure, allowing for muscle contraction and detection of spinal mobility during exercise.
Lumbar Range of Motion (cm) (change is being assessed) | Baseline and 6 weeks
  Modified- Modified Schober test For patients with low back discomfort, MMST method appears to be a good method for evaluating lumbar flexion and extension.

CONTACTS AND LOCATIONS:
Overall Officials: Farhan I Khan, Ph.D, MBA, MSc.PT, DPT, Study Director — Dow University of Health Sciences
Locations (1):
- Dow Institute of Physical Medicine and Rehabilitation, DUHS., Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No